CLINICAL TRIAL: NCT00328705
Title: D2-EPG Study: Evaluation of New Sensing Circuitry and Capture Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Collaborators: Medtronic (Industry)
Responsible Party: Cole Hannon, CRDM clinical research
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 209
Record Dates: First submitted 2006-05-19; First posted 2006-05-22 (Estimated); Last update posted 2008-02-13 (Estimated); Status verified 2008-02

CONDITIONS: Heart Diseases
Keywords: Sensing; Capture Management; Heart Failure; ICD Indication
MeSH Terms: conditions — Heart Diseases; Heart Failure | interventions — Defibrillators, Implantable

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Implantable Cardioverter Defibrillator

SUMMARY:
This is an acute, prospective, multi-center, non-randomized, investigational device exemption (IDE) clinical study.

DETAILED DESCRIPTION:
The purpose of this study is to confirm the performance of new sensing circuitry, and to confirm the performance of a Ventricular Capture Management feature in subjects with implantable cardioverter defibrillator (ICD) leads connected to an external pacemaker/defibrillator.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are scheduled for implantation or replacement of an implantable cardioverter defibrillator (ICD) or cardiac resynchronization therapy (CRT) device
* Patients must have or receive Medtronic transvenous atrial and ventricular leads in association with the scheduled device implant or replacement.

Exclusion Criteria:

* Patients who have 3rd degree heart block, as assessed by the investigator
* Patients who have a mechanical tricuspid heart valve
* Patients who have received an investigational new drug or device, or are currently enrolled in a clinical study for a new indication of an approved drug or device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2006-05; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Ventricular fibrillation (VF) detection time
Ventricular Capture Management accuracy

CONTACTS AND LOCATIONS:
Overall Officials: Cole Hannon, Study Director — Medtronic CRDM
Locations (5):
- United States (5):
  - Tampa, Florida
  - Coon Rapids, Minnesota
  - Rochester, Minnesota
  - Saint Paul, Minnesota
  - Charlotte, North Carolina